CLINICAL TRIAL: NCT03256539
Title: Napping, Sleep, Cognitive Decline and Risk of Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unexpected closure of study components -- the digital intervention (CBT-I) was no longer accessible, and alternatives were not feasible.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1K99AG056598-01 (NIH); 1K99AG056598-01 (NIH); R00AG056598 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-08-22 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Sleep; Alzheimer Disease; Cognitive Impairment; Aging; CBT
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Intervention (Experimental): Sleep treatment program (to be developed) that incorporates modified cognitive behavioral therapy for insomnia (CBT-I) and bright light therapy (BLT)
  Interventions: Behavioral: Sleep intervention
- Placebo intervention (Placebo Comparator): Placebo (quasi-desensitization) intervention for insomnia (which does not include any of the active components of CBT-I but implemented in the same frequency and duration).
  Interventions: Behavioral: Placebo intervention

INTERVENTIONS:
Behavioral: Sleep intervention — Behavioral sleep intervention program
  Arms: Sleep Intervention
Behavioral: Placebo intervention — Quasi-desensitization intervention for insomnia (which does not include any of the active components of CBT-I but implemented in the same frequency and duration)
  Arms: Placebo intervention

SUMMARY:
This study aimed to pilot test a non-pharmacological (behavioral) treatment program targeting improved cognition through improving 24-h sleep-wake cycle in people with mild cognitive impairment (MCI) or mild Alzheimer's disease. A treatment program incorporating bright light therapy and a modified cognitive behavioral therapy for insomnia will be developed to address 24-hour patterns of sleep. We will then pilot test its feasibility and explore its preliminary effects on improving sleep/napping and cognition in patients with MCI or mild Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* Memory complaints verified by an informant
* Clinical diagnosis of mild cognitive impairment (MCI) or mild Alzheimer's Disease
* General cognitive performance sufficiently persevered such that a diagnosis of Alzheimer's disease cannot be made by the site physician
* No evidence (CT or MRI scans within 12 months prior to screening) of infection, infarction, or other focal lesions and no clinical symptoms suggestive of intervening neurological disease
* Adequate visual and auditory acuity to allow neuropsychological testing
* Meets International Classification of Sleep Disorders-2nd edition (ICSD-2) criteria for insomnia or circadian rhythm disorders, or shows actigraphy evidence of sleep disturbances and excessive napping

Exclusion Criteria:

* Any major neurologic disease other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, multiple sclerosis, seizure disorder, Huntington's disease, brain tumor or history of significant head trauma
* Any comorbid psychiatric conditions or severe personality disorder within the past 2 years (by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition), such as major depression, bipolar disorder, schizophrenia and other psychotic features
* Any uncontrolled medical conditions or systemic illness that might lead to difficulty complying with the study protocol
* History of alcohol or substance abuse within the past 2 years
* Any inadequately treated primary or secondary sleep disorder (due to medical conditions) that might confound the association

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Leng, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep Intervention: An FDA-authorized prescription digital cognitive behavioral therapy for insomnia (CBT-I) therapeutic treatment
- Placebo Intervention: Placebo (quasi-desensitization) intervention for insomnia (which does not include any of the active components of CBT-I but implements in the same frequency and duration).
Period: Overall Study
Arm/Group | Sleep Intervention | Placebo Intervention
Started | 8 | 7
Completed | 0 | 0
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Unexpected closure of study components | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Intervention | Placebo Intervention | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (5.15) | 74.1 (4.81) | 74.93 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) ranges from 0-21, with higher scores indicating worse sleep quality.
  units on a scale | 9.88 (3.18) | 11.4 (3.51) | 10.6 (3.31)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) ranges from 0-28, with higher scores indicating worse insomnia symptoms. Scoring is as follows: 0 - 7 No clinically significant insomnia; 8 - 14 Subthreshold insomnia; 15 - 21 Clinical insomnia (moderate severity); 22 - 28 Clinical insomnia (severe).
  units on a scale | 16.8 (5.52) | 15.2 (4.90) | 16.03 (5.11)
Quick Dementia Rating System (QDRS) Category [Count of Participants; unit: Participants]
  Mild cognitive impairment | 4 | 4 | 8
  Mild dementia | 4 | 3 | 7
STOP-BANG sleep apnea scale [Count of Participants; unit: Participants] — The STOP-BANG sleep apnea scale assesses risk of sleep apnea and consists of eight yes or no questions. Scoring is as follows: Low Risk: Yes to 0 - 2 questions; Intermediate Risk: Yes to 3 - 4 questions; High Risk: Yes to 5 - 8 questions.
  Participants
    High risk | 1 | 0 | 1
    Intermediate risk | 5 | 1 | 6
    Low risk | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled to the Study
Time Frame: Up to 24 weeks following study initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Intervention | Placebo Intervention
Number analyzed (Participants) | 8 | 7
Participants | 8 | 7

2. Primary Outcome: Number of Participants That Complete the Study
Time Frame: Through study completion, up to 34 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points.
Arm/Group | Sleep Intervention | Placebo Intervention
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Sleep as Assessed by Actigraphy
Description: Week-long measurement using wrist actigraphy
Time Frame: Through study completion, up to 34 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points.
Arm/Group | Sleep Intervention | Placebo Intervention
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cognitive Function Assessed by Standard Neurocognitive Battery
Time Frame: Through study completion, up to 34 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points.
Arm/Group | Sleep Intervention | Placebo Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Sleep Intervention | Placebo Intervention
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT03256539/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT03256539/SAP_001.pdf
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT03256539/ICF_002.pdf